CLINICAL TRIAL: NCT00170872
Title: A 6 Week, Multicenter, Open-label Trial to Evaluate the Safety, Tolerability and Efficacy of Lumiracoxib 200mg o.d. in Patients With Primary Knee Osteoarthritis or Rheumatoid Arthritis
Brief Title: 6 Week Open-label Trial With Lumiracoxib 200mg o.d. in Primary Knee Osteoarthritis or Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCOX189A2365
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis
Keywords: Osteoarthritis; Rheumatoid Arthritis; Cox-2; lumiracoxib
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid | interventions — lumiracoxib

INTERVENTIONS:
Drug: Lumiracoxib

SUMMARY:
This study tested the safety, tolerability and efficacy of lumiracoxib - a COX-2 inhibitor- in patients with primary knee osteoarthritis or rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Requirement of regular NSAID therapy
* With primary osteoarthritis of the target knee (by ACR Criteria) or with a diagnosis of rheumatoid arthritis (by ACR Criteria)

Exclusion Criteria:

* Evidence of active ulceration of the UGI tract within 6 months prior to the screening visit or history of active bleeding of the UGI tract within the previous 5 years. As well as with pyloric or duodenal obstruction or with history of gastrointestinal parasites.
* History of cardiac and cerebral thrombotic/ischemic diseases and/or events
* Patients taking additional NSAIDs (including COX-2 inhibitors) during the course of the study.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 135
Dates: Start 2004-11; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Assess safety and tolerability profile of lumiracoxib in comparison to baseline

SECONDARY OUTCOMES:
Demonstrate that lumiracoxib 200mg o.d. is effective in treating OA and pain due to RA with respect to overall OA/ RA pain intensity on a 0-100 mm Visual Analog Scale (VAS) after 6 weeks of treatment in comparison to baseline
Assess efficacy of lumiracoxib compared to baseline with respect to a) overall OA/ RA pain intensity b) patient's and physician's global assessment of disease activity c) patient functional status
Use of rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Chair — Sponsor GmbH